CLINICAL TRIAL: NCT06016777
Title: Optimization of Perioperative Analgesia Protocol for Uniportal Video-assisted Thoracoscopic Surgery: a Randomized Controlled Trial
Brief Title: Optimization of Perioperative Analgesia Protocol for Uniportal Video-assisted Thoracoscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Li Fang Wang, attending doctor, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ChinaJapanFHAnesth2
Record Dates: First submitted 2023-08-14; First posted 2023-08-30 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Uniportal Video-assisted Thoracic Surgery
Keywords: fast-track; Enhanced Recovery After Surgery; uniportal video-assisted thoracoscopic surgery; randomized controlled trial; thoracoscopic; ultrasonic guidance; paravertebral block; erector spinal block

STUDY DESIGN:
Intervention Model Description: This will be a parallel-group, single-blind, randomized controlled trial. Patients are expected to be enrolled in the trial within 8 months. Participants will be randomly assigned to one of the three groups: ultrasound-guided paravertebral block (PVB+PCIA group), ultrasound-guided erector spinae block(ESB+PCIA group) , or intravenous patient-controlled analgesia pump group (PCIA group). Different nerve block operation schemes will be used in different groups.Except for different nerve block schemes, all the participants will have the same methods and choices of medicine for other kinds of rescue analgesia regimens.The participants and the follow-up evaluation doctors are not aware of the group assignment, and the surgeon and anesthesiologist will not know the grouping code until the beginning of the surgery. In this way, the analgesic effect of each subject can be fairly evaluated.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients will be grouped by block randomization method (1:1:1) by a researcher who is unaware of the meaning of the group code. Patients will be stratified by ID numbers with a block of 6. Within each block, random sequences between 0 and 1 are generated. The group code (A, B or C) will be defined as the remainder of the serial number divided by three. The group code will be put in a light-proof envelope. Patients with the envelope will be transferred to the OR, unaware of the group assignment throughout the study. After induction, the anesthesiologist opens the light-proof envelope and get the group code. Group codes will be recorded in the CRF table with the cards destroyed. Only the principal investigator and the anesthesiologists know the intervention represented by the group code. The anesthesiologists will not involve in postoperative follow-ups or data collection. Neither doctors in charge of postoperative follow-ups nor the statisticians will know the specific interventions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PVB+PCIA group (Experimental)
  Interventions: Procedure: Ultrasound-guided paraspinal block and patient-controlled intravenous analgesia pump; Procedure: Patient-controlled intravenous analgesia pump
- ESB+PCIA group (Experimental)
  Interventions: Procedure: Ultrasound-guided erector spinal block and patient-controlled intravenous analgesia pump; Procedure: Patient-controlled intravenous analgesia pump
- PCIA group (Active Comparator)
  Interventions: Procedure: Patient-controlled intravenous analgesia pump

INTERVENTIONS:
Procedure: Ultrasound-guided paraspinal block and patient-controlled intravenous analgesia pump — Patients in this group will receive ultrasound-guided paraspinal block with 0.3% ropivacaine and 5mg dexamethasone in total of 20mL saline at T5 level on the operative side. Patients in all the groups will be treated with PCIA after surgery. PCIA with sufentanil will be applied to all participants, with background infusion at 1.8μg/hour, and total dosage <5μg/hour.
  Arms: PVB+PCIA group
Procedure: Ultrasound-guided erector spinal block and patient-controlled intravenous analgesia pump — Patients in this group will receive ultrasound-guided erector spinal block with 0.3% ropivacaine and 5mg dexamethasone in total of 20mL saline at T5 level on the operative side. Patients in all the groups will be treated with PCIA after surgery. PCIA with sufentanil will be applied to all participants, with background infusion at 1.8μg/hour, and total dosage <5μg/hour.
  Arms: ESB+PCIA group
Procedure: Patient-controlled intravenous analgesia pump — Patients in this group will not receive regional block. Patients in all the groups will be treated with PCIA after surgery. PCIA with sufentanil will be applied to all participants, with background infusion at 1.8μg/hour, and total dosage <5μg/hour.

SUMMARY:
Trial design Despite video-assisted thoracic technology and procedure specific postoperative pain management (PROSPECT) have been promoted through recent years, thoracic surgery is still considered to be one of the most painful of surgical procedures. This study aims to optimize these conditions according to different perioperative analgesic modes recommended at present. This will be a single-blind randomized study to investigate the optimal analgesic effect of thoracic paravertebral block (TPB), erector spinae block (ESB), or sufentanil patient controlled intravenous analgesia (PCIA) for uniportal video-assisted thoracoscopic surgery (uVATS) and using minimally invasive drainage.

Methods One-hundred and two patients undergoing uVATS will be enrolled. Patients will be randomly assigned to PVB group (20mL 0.3% ropivacaine with dexamethasone), ESB group (20mL 0.3% ropivacaine with dexamethasone) or CON group. PCIA with sufentanil will be provided to all patients after surgery. Primary outcome will be total opioid consumption from the end of the surgery to the time of discharge. Secondary outcomes consist of postoperative pain score, postoperative chronic pain, both at rest and during coughing, sensations of touch and pain on the chest wall, non-opioid analgesic drug use, length of stay (LOS), ambulation time, total cost of hospitalization and long-term postoperative analgesia. Adverse reaction to analgesics and adverse event related to regional block will also be recorded.

Ethics and dissenmination This study is approved by the Ethics Committee of China-Japan Friendship Hospital (ID 2022-KY-127-1). The results will be published in peer-reviewed journals.

Key words: fast-track; Enhanced Recovery After Surgery; uniportal video-assisted thoracoscopic surgery; randomized controlled trial; thoracoscopic; ultrasonic guidance; paravertebral block; erector spinal block

DETAILED DESCRIPTION:
This is a prospective, randomized controlled study. Patients who are scheduled for elective uniportal thoracoscopic surgery in our hospital will be enrolled. Patients will be randomly assigned to one of the three groups: ultrasound-guided paravertebral block, ultrasound-guided erector spinae block, or intravenous patient-controlled analgesia pump group. Different nerve block operation schemes will be used in different groups.

In any of the three groups, general anesthesia will be performed according to the standard, and multi-mode analgesic treatment will be appied as the combination of NSAIDs analgesics, opioid analgesics, and postoperative rescue analgesic treatment. Participants will be followed up at 1, 4, 12, 18 hours, on 1, 2, 3, 4, 7 days, and in 1, 2, 3, 4, 6 months after surgery. At each follow-up visit, rest and cough pain level will be recorded, and sense of touch and pain in the chest will be examined. Additional analgesic treatment will be given if necessary.

Comparisons of the postoperative analgesic use, cough and rest pain, ambulation time, length of hospital stay, and hospital costs will be made in the three groups.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years
2. ASA I-IIa
3. Early stage lung cancer or intrathoracic tissue biopsy, suitable for elective uVATSb
4. Informed consent obtained

Exclusion Criteria:

1. ASA≥III
2. History of intrathoracic or chest wall surgery
3. Chronic pain
4. Pre-operative analgesic medication use
5. NSAIDsc contraindications: aspirin asthma, allergic to NSAIDs, peptic ulcer, liver and kidney insufficiency, high risk of thrombotic events
6. Active autoimmune disease
7. Allergic to local anesthetics
8. Severe coagulation dysfunction, contraindicated for nerve block
9. Soft tissue infections of the chest wall

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
total opioid consumption | up to 6 months, total opioid use from postoperative period till the discontinuation of surgery-related therapy.
  total opioid (morphine equivalent/body weight) consumption from the end of the surgery to the time of discharge.

SECONDARY OUTCOMES:
postoperative pain score assessed by Visual Analogue Scale VAS (1-10) | from the time at the end of surgery to 24 weeks after surgery
  rest and cough pain
postoperative pain score assessed by Numeric Rating Scales, NRS (1-10) | from the time at the end of surgery to 24 weeks after surgery
  rest and cough pain
sensations of touch on the chest wall | from the time at the end of surgery to 24 weeks after surgery
  difference in tactile sense on bilateral chest-wall. Tactile sensation and cold sensation will be measured at four points (<3cm near the incision, and on the other side on the symmetrical chest wall, and at the point of bilateral mid-clavicular-costal arch) with an alcohol-stained cotton swab
non-opioid analgesic drug use | from the time at the end of surgery to 24 weeks after surgery
  number of patients with long-term (≥3 days) use of non-opioid analgesic drug
length of stay (LOS) | up to 1 month, LOS is the amount of days the patient spends in the hospital, determined by subtracting the date of admission from the date of discharge
  days of hospital stay
ambulation time | up to 1 month, ambulation time is the time the patient first ambulated following the surgical procedure
  first time of successful activity off bed, the time between the end of surgery to the time of the first successful ambulation
total cost of hospitalization | up to 1 month, total charges settled on the day of discharge
  the in-patients costs total cost of hospitalization=medication cost + hospitalization cost + nursing cost + delay compensation
long-term postoperative analgesia | from the time at the end of surgery to 24 weeks after surgery
  number of patient who needs long-term postoperative analgesia (≥3 days after discharge)
adverse events | from the time at the end of surgery to 24 weeks after surgery
  Adverse reactions such as dizziness, nausea, vomiting, drowsiness, dyspnea, fatigue, constipation and urinary retention were recorded in detail
chest tube removal time | from the time at the end of surgery to 24 weeks after surgery
  The time from surgery to removal of the chest drainage tube

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Rong ZHANG, Doctor, Study Director — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Security cameras are set up next to both the computer and the cabinet for data storage. The surveillance video will be available only to medical staff and the principal investigator. Access to data will be restricted to authorized personnel, including ethics committee directors, principal investigator and authorized personnel. Access to paper documents as well as electronic data must be registered, with the name of operator and detailed reasons recorded.
  The results and conclusions of our research will be reported to all the participants, research team, and the public in peer-reviewed journal. The investigators will try to put forward the existing guidelines to further optimization of perioperative anesthesia and analgesia protocol for small-incision thoracic surgery and optimized drainage tube strategy.

REFERENCES:
- [Derived] Wang LF, Qi F, Feng HX, Shi YH, Li Y, Zheng MT, Bu T, Li WX, Zhang ZR. Risk and benefit analysis of single-shot nerve block for postoperative analgesia for uniportal video-assisted thoracic surgery (uVATS): a randomized controlled trial. BMC Anesthesiol. 2025 Feb 12;25(1):68. doi: 10.1186/s12871-025-02955-w. PMID 39939956
- [Derived] Wang LF, Feng HX, Shi YH, Li Y, Zheng MT, Bu T, Zhang ZR. Protocol for a randomised controlled trial: optimisation of perioperative analgesia protocol for uniportal video-assisted thoracoscopic surgery. BMJ Open. 2024 Apr 2;14(4):e079434. doi: 10.1136/bmjopen-2023-079434. PMID 38569709